CLINICAL TRIAL: NCT01532193
Title: A Randomized Controlled Trial Evaluation the Effect of Low Oxygen Tension on the Pregnancy Rate After Day 3 Embryo Transfer in an Egg Donation Programme.
Brief Title: The Effect of Embryo Culture Under Low Oxygen Tension on Pregnancy Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Maria Jose Delossantos, Dr. Maria Jose Delossantos, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0903-C-059-MJ
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Low Oxygen Tension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hipoxia (Experimental): The low oxygen tension group
  Interventions: Other: Decreased oxygen concentration
- Control group (No Intervention): Conventional culture conditions

INTERVENTIONS:
Other: Decreased oxygen concentration — The oxygen concentration is decreased during the "in Vitro" embryo culture.
  Arms: Hipoxia

SUMMARY:
This study will determine whether the use of low oxygen tension during "in vitro" embryo culture may increase the pregnancy rates in women undergoing egg donation.

DETAILED DESCRIPTION:
As far as oxygen (O2) tension is concerned, both oocytes and embryos from different mammalian species included the human are normally surrounded by values which are much less than half of atmospheric O2, ranging from high (8.7% O2) in the rabbit oviduct, rabbit and hamster uterus, to as low as 11 mm Hg (1.5% O2) in the monkey uterus. Even in the preovulatory follicle, oocytes are bathed within follicular fluids containing oxygen that range from > 1 to 5.5 % The aim of this study was to evaluate the impact the effect of low oxygen tension after day-3 embryo transfer in our egg donation programme on pregnancy and implantation rates.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25-45 years of age;
* In good mental and physical health;
* First or second of egg-recipient treatment;
* Embryo transfer on Day 3.
* One to three embryos will be transferred.
* BMI between 18-25 kg/m2.

Exclusion Criteria:

* Uterine pathology or hydrosalpinx
* Recurrent miscarriage
* No chronic illnesses

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rates per cycle | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Ivi Valencia, Valencia, Spain

REFERENCES:
- [Derived] Rendon Abad M, Serra V, Gamiz P, de Los Santos JM, Remohi J, Navarro AT, de Los Santos MJ. The influence of oxygen concentration during embryo culture on obstetric and neonatal outcomes: a secondary analysis of a randomized controlled trial. Hum Reprod. 2020 Sep 1;35(9):2017-2025. doi: 10.1093/humrep/deaa152. PMID 32772073